CLINICAL TRIAL: NCT01756040
Title: Gut Permeability in Very Low Birth Weight Infants
Brief Title: Intestinal Permeability in Preterm Infants
Acronym: IPPI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Rose Viscardi, University of Maryland, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HP-00049647
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Prematurity; Intestinal Permeability
Keywords: intestinal permeability; preterm infants; dual sugar test; intestinal microbiota
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lactulose - rhamnose solution (Other): Preterm Infants age 24-32 weeks gestation
  Interventions: Drug: Lactulose -rhamnose solution

INTERVENTIONS:
Drug: Lactulose -rhamnose solution — Measurement of intestinal permeability by use of mon- digestible sugars known not to cross the intestinal barrier in normal healthy intestinal tissue
  Other Names: dual sugar solution

SUMMARY:
Necrotizing enterocolitis (NEC) is a life-threatening, gastrointestinal emergency characterized by increased intestinal permeability, affects approximately 7 to 10% of infants <1500 g birthweight, and typically occurs within 7 to 14 days of birth. Mortality is as high as 30-50%. Prematurity is the greatest risk factor for the development of NEC due to the physiological immaturity of the gastrointestinal tract and altered or abnormal gut microbiota. Several studies have demonstrated that the initiation of an intense systemic and local inflammatory cascade leads to intestinal necrosis. The human intestine is lined by a single layer of cells exquisitely responsive to multiple stimuli and is populated by a complex climax community of microbial partners. Under normal circumstances, these intestinal cells form a tight but selective barrier to "friends and foes": microbes and most environmental substances are held at bay, but nutrients are absorbed efficiently. Epithelial barrier integrity is itself dynamic and matures over time starting soon after birth, though the mechanisms regulating dynamic permeability are poorly understood. Low birth weight, prematurity, and early postnatal age are associated with a leaky gut. Although intestinal permeability is higher at birth in preterm than term infants, there is usually rapid maturation of the intestinal barrier over the first few days of life in both populations. The investigators hypothesize that increased levels of measures of intestinal permeability (urine lactulose/rhamnose (LA/Rh), and fecal alpha1- antitrypsin will identify infants at high risk for NEC and that intestinal probiotic strains will be associated with intestinal barrier maturation. The purpose of the study is to determine whether clinical factors in combination with non-invasive stool test such as antitrypsin (A1AT) and microbiota composition profile are associated with intestinal permeability determined by excretion of non-metabolized sugar probes in urine (LA/Rh ratio). These studies may lead to a non-invasive screening test to identify preterm infants at risk for NEC.

DETAILED DESCRIPTION:
The proposed study will evaluate the intestinal permeability measured by the urinary La/Rh ratio at one timepoint between d7-10 of life in 200 preterm infants 24-32 weeks gestation in preparation for a future study of probiotics to improve intestinal permeability in this population.

Primary Objective: To estimate mean and variance in IP measured by urinary Lactulose/Rhamnose ratio at 7-10d of life in neonates born between 24 and 32 weeks of gestational age.

Secondary Objectives

1) To assess stool microbiome characteristics in association with intestinal permeability in preterm infants measured by the urinary lactulose/rhamnose ratio.

ELIGIBILITY:
Inclusion Criteria:

* <5 days
* Gestational age 24-32 weeks

Exclusion criteria:

* Nonviable or planned withdrawal of care
* Significant GI dysfunction (e.g. heme-positive stools, abdominal distension (girth >2 cm baseline), or bilious emesis/aspirates.
* Triplet or higher order multiple
* Severe asphyxia
* Lethal chromosome abnormalities
* Cyanotic congenital heart disease
* Intestinal atresia or perforation
* Abdominal wall defects
* Known galactosemia or other galactose intolerance

Max Age: 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Fasano, MD, Principal Investigator — Massachusetts General Hospital; Rose M Viscardi, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fasano A. Physiological, pathological, and therapeutic implications of zonulin-mediated intestinal barrier modulation: living life on the edge of the wall. Am J Pathol. 2008 Nov;173(5):1243-52. doi: 10.2353/ajpath.2008.080192. Epub 2008 Oct 2. PMID 18832585
- [Background] Bjarnason I. Intestinal permeability. Gut. 1994 Jan;35(1 Suppl):S18-22. doi: 10.1136/gut.35.1_suppl.s18. PMID 8125384
- [Background] van Wijck K, Bessems BA, van Eijk HM, Buurman WA, Dejong CH, Lenaerts K. Polyethylene glycol versus dual sugar assay for gastrointestinal permeability analysis: is it time to choose? Clin Exp Gastroenterol. 2012;5:139-50. doi: 10.2147/CEG.S31799. Epub 2012 Jul 19. PMID 22888267
- [Background] van Wijck K, Verlinden TJ, van Eijk HM, Dekker J, Buurman WA, Dejong CH, Lenaerts K. Novel multi-sugar assay for site-specific gastrointestinal permeability analysis: a randomized controlled crossover trial. Clin Nutr. 2013 Apr;32(2):245-51. doi: 10.1016/j.clnu.2012.06.014. Epub 2012 Aug 11. PMID 22892368
- [Background] Beach RC, Menzies IS, Clayden GS, Scopes JW. Gastrointestinal permeability changes in the preterm neonate. Arch Dis Child. 1982 Feb;57(2):141-5. doi: 10.1136/adc.57.2.141. PMID 7065710
- [Background] Piena-Spoel M, Albers MJ, ten Kate J, Tibboel D. Intestinal permeability in newborns with necrotizing enterocolitis and controls: Does the sugar absorption test provide guidelines for the time to (re-)introduce enteral nutrition? J Pediatr Surg. 2001 Apr;36(4):587-92. doi: 10.1053/jpsu.2001.22288. PMID 11283883
- [Background] Rouwet EV, Heineman E, Buurman WA, ter Riet G, Ramsay G, Blanco CE. Intestinal permeability and carrier-mediated monosaccharide absorption in preterm neonates during the early postnatal period. Pediatr Res. 2002 Jan;51(1):64-70. doi: 10.1203/00006450-200201000-00012. PMID 11756641
- [Background] Albers MJ, Steyerberg EW, Hazebroek FW, Mourik M, Borsboom GJ, Rietveld T, Huijmans JG, Tibboel D. Glutamine supplementation of parenteral nutrition does not improve intestinal permeability, nitrogen balance, or outcome in newborns and infants undergoing digestive-tract surgery: results from a double-blind, randomized, controlled trial. Ann Surg. 2005 Apr;241(4):599-606. doi: 10.1097/01.sla.0000157270.24991.71. PMID 15798461
- [Background] Piena M, Albers MJ, Van Haard PM, Gischler S, Tibboel D. Introduction of enteral feeding in neonates on extracorporeal membrane oxygenation after evaluation of intestinal permeability changes. J Pediatr Surg. 1998 Jan;33(1):30-4. doi: 10.1016/s0022-3468(98)90355-4. PMID 9473094
- [Background] Malagon I, Onkenhout W, Klok M, van der Poel PF, Bovill JG, Hazekamp MG. Gut permeability in neonates after a stage 1 Norwood procedure. Pediatr Crit Care Med. 2005 Sep;6(5):547-9. doi: 10.1097/01.pcc.0000175990.72753.97. PMID 16148815
- [Background] Noone C, Menzies IS, Banatvala JE, Scopes JW. Intestinal permeability and lactose hydrolysis in human rotaviral gastroenteritis assessed simultaneously by non-invasive differential sugar permeation. Eur J Clin Invest. 1986 Jun;16(3):217-25. doi: 10.1111/j.1365-2362.1986.tb01332.x. PMID 3089818
- [Background] van Elburg RM, Fetter WP, Bunkers CM, Heymans HS. Intestinal permeability in relation to birth weight and gestational and postnatal age. Arch Dis Child Fetal Neonatal Ed. 2003 Jan;88(1):F52-5. doi: 10.1136/fn.88.1.f52. PMID 12496227
- [Background] Catassi C, Bonucci A, Coppa GV, Carlucci A, Giorgi PL. Intestinal permeability changes during the first month: effect of natural versus artificial feeding. J Pediatr Gastroenterol Nutr. 1995 Nov;21(4):383-6. doi: 10.1097/00005176-199511000-00003. PMID 8583288
- [Derived] Roskes L, Chamzas A, Ma B, Medina AE, Gopalakrishnan M, Viscardi RM, Sundararajan S. Early human milk feeding: Relationship to intestinal barrier maturation and postnatal growth. Pediatr Res. 2025 May;97(6):2065-2073. doi: 10.1038/s41390-024-03622-5. Epub 2024 Oct 14. PMID 39397156
- [Derived] Mahdally SM, Izquierdo M, Viscardi RM, Magder LS, Crowley HM, Bafford AC, Drachenberg CB, Farfan MJ, Fasano A, Sztein MB, Salerno-Goncalves R. Secretory-IgA binding to intestinal microbiota attenuates inflammatory reactions as the intestinal barrier of preterm infants matures. Clin Exp Immunol. 2023 Oct 13;213(3):339-356. doi: 10.1093/cei/uxad042. PMID 37070830
- [Derived] Saleem B, Okogbule-Wonodi AC, Fasano A, Magder LS, Ravel J, Kapoor S, Viscardi RM. Intestinal Barrier Maturation in Very Low Birthweight Infants: Relationship to Feeding and Antibiotic Exposure. J Pediatr. 2017 Apr;183:31-36.e1. doi: 10.1016/j.jpeds.2017.01.013. Epub 2017 Jan 31. PMID 28159311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants born 24-32 weeks gestation were enrolled at a level IV Neonatal Intensive Care Unit at the University of Maryland Medical Center in the intestinal permeability study during 2 enrollment periods [Cohort 1(April 15, 2013-October 15, 2014) (N=44)] and [Cohort 2 (October 15, 2018-June 11, 2021) (N=167)].
Pre-assignment Details: Parental consent was obtained for 214 infants, but parents of three infants withdrew consent prior to receipt of the sugar probe (lactulose/rhamnose) dose. Two infants died after consent, but before receiving the sugar probe dose. Seven infants were not dosed due to feeding intolerance (N=4), spontaneous intestinal perforation (N=2), transfer/discharge prior to dosing day (N=1). The remaining 201 enrolled infants received at least 1 dose of the sugar probe.
Period: IP in Preterm Infants: Cohort 1
Arm/Group | Lactulose - Rhamnose Solution
Started | 44
Completed | 43
Not Completed | 1
Not completed — Death | 1
Period: IP in Preterm Infants: Cohort 2
Arm/Group | Lactulose - Rhamnose Solution
Started | 167
Completed | 158
Not Completed | 9
Not completed — Death | 1
Not completed — did not receive sugar probe dose | 8

BASELINE CHARACTERISTICS:
Population: The baseline population is the number of infants enrolled in the study.
Arm/Group | Lactulose - Rhamnose Solution
Number analyzed (Participants) | 211
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 211
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 1.93 (1.08)
Age, Customized [Count of Participants; unit: Participants]
  Gestational age: Gestational age 24wk 0d-28wk6d | 63
  Gestational age: Gestational age 29wk 0 d- 32 wk 6d | 148
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 204
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 123
  White | 72
  More than one race | 2
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 211
Birthweight [Count of Participants; unit: Participants]
  <1000 gm BW | 53
  ≥1000 gm BW | 158

OUTCOME MEASURES:

1. Primary Outcome: Intestinal Permeability
Description: Intestinal Permeability measured by urinary excretion of orally administered lactulose/rhamnose (La/Rh ratio)
Time Frame: 7-10 days postnatal
Population: Study participants who had lactulose/rhamnose sugar solution administered between 7-10 days postnatal age and urine collected over 4 hours that was measured for lactulose/rhamnose concentration by HPLC.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Gestational Age <29 wk: Preterm Infants age 24wk 0 d-28 wk 6 d gestation
- Gestational Age ≥29 Weeks: Participants with gestational age at birth 29 wk 0 d to 32 wk 6 d
Arm/Group | Gestational Age <29 wk | Gestational Age ≥29 Weeks
Number analyzed (Participants) | 55 | 134
ratio | 0.0731 (0.0076) | 0.0720 (0.0078)
Statistical Analysis 1: Comparison: Gestational Age <29 wk vs Gestational Age ≥29 Weeks; We hypothesized that intestinal permeability as measured by urinary lactulose/rhamnose ratio would be higher in the lower gestational age (<29 weeks) compared to the more mature infants (≥29 weeks gestation) at postnatal age 7-10 days; Test type: Other; p = 0.932, t-test, 2 sided — not adjusted for multiple comparisons. The a priori threshold for statistical significance was <0.05

2. Secondary Outcome: Stool Alpha-1 Antitrypsin
Description: Stool alpha-1 antitrypsin concentrations
Time Frame: 7-10 days postnatal
Population: Infants at 7-10 days of age in the first cohort who had stool collected on the same day as urinary IP measurement that was assayed by ELISA for A1AT concentration.
Measure: Mean (Standard Deviation); unit: µg/ml
Groups:
- Low Intestinal Permeability (IP) Group: Normal intestinal barrier function or low IP was defined as urinary lactulose/rhamnose ratio ≤0.05
- High IP Group: Infants with high intestinal permeability (indicator of impaired intestinal barrier function) as measured by urinary lactulose/rhamnose ratio >0.05
Arm/Group | Low Intestinal Permeability (IP) Group | High IP Group
Number analyzed (Participants) | 6 | 7
µg/ml | 359.5 (137.0) | 1285.3 (802.3)
Statistical Analysis 1: Comparison: Low Intestinal Permeability (IP) Group vs High IP Group; We hypothesized that stool A1AT would be higher in infants with high IP as measured by urinary La/Rh compared to those with low IP; Test type: Other; p = 0.316, t-test, 2 sided

3. Secondary Outcome: Stool Microbiota Relative Abundance
Description: Relative abundance (%) Clostridiales species
Time Frame: 7-10 days postnatal
Population: Infants who had both urinary La/Rh ratio and stool Clostridiales abundance determined
Measure: Median (Inter-Quartile Range); unit: percentage of Clostridiales in stool
Arm/Group | Low Intestinal Permeability (IP) Group | High IP Group
Number analyzed (Participants) | 43 | 36
percentage of Clostridiales in stool | 6.52 [0.108 to 15.68] | 0.07 [0.003 to 0.605]
Statistical Analysis 1: Comparison: Low Intestinal Permeability (IP) Group vs High IP Group; Test type: Other; p = 0.011, Bayesian goodness of fit — The significance value was estimated using Bayesian goodness-of-fit p-value to assess the significance of the association of the relative abundance of Clostridiales and IP categories. P value <0.05 was considered significant

4. Secondary Outcome: Breastmilk Feeding Duration Prior to La/Rh Measurement
Description: Number of days breast milk feeding prior to La/Rh measurement between d7-10 days of age.
Time Frame: 7-10 days postnatal
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Low Intestinal Permeability (IP) Group | High IP Group
Number analyzed (Participants) | 76 | 50
days | 7.02 (1.38) | 6.1 (1.96)
Statistical Analysis 1: Comparison: Low Intestinal Permeability (IP) Group vs High IP Group; We hypothesized that infants with normal barrier function (La/Rh ratio ≤0.05) would have been fed breastmilk for longer duration than infants with impaired barrier function (La/Rh>0.05); Test type: Other; p = 0.0023, t-test, 2 sided

5. Other Pre Specified Outcome: Occurrence of Necrotizing Enterocolitis
Description: Frequency of ≥ Stage 2 Necrotizing enterocolitis
Time Frame: 0-28 days postnatal
Population: Infants who had urinary La/Rh measured between 7-10 days of age (total N=189)
Measure: Count of Participants; unit: Participants
Arm/Group | Low Intestinal Permeability (IP) Group | High IP Group
Number analyzed (Participants) | 105 | 84
Participants | 0 | 0
Statistical Analysis 1: Comparison: Low Intestinal Permeability (IP) Group vs High IP Group; Test type: Other; p = 1.0, Chi-squared

6. Other Pre Specified Outcome: Percent Participants Exposed to Antibiotics Prior to La/Rh Measurement
Description: Percent of participants with antibiotic exposure prior to La/Rh measurement
Time Frame: 7-10 days postnatal
Population: Study participants who had urinary La/Rh ratio measured on postnatal day 7-10.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Intestinal Permeability (IP) Group | High IP Group
Number analyzed (Participants) | 105 | 84
Participants | 79 | 67
Statistical Analysis 1: Comparison: Low Intestinal Permeability (IP) Group vs High IP Group; Test type: Other; p = 0.461, Chi-squared — A priori threshold <0.05

7. Other Pre Specified Outcome: Postnatal Age Full Feeds Reached
Description: Postnatal age when all nutrition is provided by enteral feeds
Time Frame: 0-100 days postnatal
Population: Study participants who had urinary La/Rh ratio measured between 7-10 days of age.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Low Intestinal Permeability (IP) Group | High IP Group
Number analyzed (Participants) | 105 | 84
days | 11.46 (5.04) | 22.02 (45.5)
Statistical Analysis 1: Comparison: Low Intestinal Permeability (IP) Group vs High IP Group; We hypothesized that infants with impaired barrier function as measured by high urinary La/Rh (>0.05) ratio at 7-10 days of age would require longer time to reach full enteral feedings than infants with normal barrier function (La/Rh≤0.05); Test type: Other; p = 0.019, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Birth- 28 days of life.
Description: Adverse events were collected daily for participants.
Arm/Group | Lactulose - Rhamnose Solution
All-Cause Mortality (participants affected / at risk) | 2/211
Serious Adverse Events (participants affected / at risk) | 22/211
Other Adverse Events (participants affected / at risk) | 32/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactulose - Rhamnose Solution (N=211)
Progressive hydrocephalus (Nervous system disorders) | 1 (1)
Intraventricular hemorrhage, Grade IV (Nervous system disorders) | 2 (2)
Intraventricular hemorrhage, Grade III (Nervous system disorders) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary interstitial emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Worsening respiratory status (Respiratory, thoracic and mediastinal disorders) | 3 (3) — worsening respiratory status requiring increased support such as intubation and mechanical ventilation
patent ductus arteriosus (Cardiac disorders) | 4 (4) — patent ductus arteriosus that was treated with medication (e.g. indomethacin)
Spontaneous intestinal perforation (Gastrointestinal disorders) | 1 (1)
direct hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) — Direct conjugated bilirubin >2.0 mg/dL
sepsis (Infections and infestations) | 4 (4) — culture-confirmed bloodstream infection (sepsis)
Urinary tract infection (Infections and infestations) | 1 (1) — Culture-confirmed urinary tract infection
pleocytosis (Blood and lymphatic system disorders) | 1 (1) — Elevated WBC count (severity IV)
neutropenia (Blood and lymphatic system disorders) | 1 (1) — low white blood cell count <2000
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) — Serum calcium >12.2 meq/L
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) — Serum potassium ≥6.9
metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) — Serum bicarbonate <15 meq/L
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactulose - Rhamnose Solution (N=211)
Vomiting (Gastrointestinal disorders) | 10 (10) — vomiting <5 episodes/day
low serum bicarbonate (Blood and lymphatic system disorders) | 23 (23) — Serum bicarbonate 15-21 meq/L
hyperkalemia (Metabolism and nutrition disorders) | 14 (14) — Serum potassium >5.5 and <6.9
Elevated BUN (Metabolism and nutrition disorders) | 11 (11) — Blood urea nitrogen (BUN) >27 and <59 meq/L
anemia (Blood and lymphatic system disorders) | 11 (11) — hematocrit <35 and >25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT01756040/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT01756040/ICF_001.pdf